CLINICAL TRIAL: NCT04680585
Title: Reproductive Mental Health of Ontario Virtual Intervention Network (MOVIN): A Pilot Randomized Controlled Trial
Brief Title: MOVIN Pilot Randomized Controlled Trial
Acronym: MOVIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Principal Investigator, Simone Vigod, Chief, Department of Psychiatry, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2020-0054-B
Record Dates: First submitted 2020-12-07; First posted 2020-12-23 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Depression, Postpartum
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (Other): Access to online resources and educational materials about general mental health, maternal mental health, depression and anxiety in the pregnancy and postpartum period, and an up-to-date listing of treatment services available in Ontario. These resources are maintained by the MOVIN study team.
  Interventions: Other: Enhanced Usual Care
- MOVIN (Experimental): Enhanced Usual Care plus MOVIN Care Platform. The MOVIN Care Platform is virtual collaborative care intervention with a stepped care approach in which a care coordinator directs participants to one or more evidence-based virtual interventions as appropriate.
  Interventions: Other: Enhanced Usual Care; Other: MOVIN Care Platform

INTERVENTIONS:
Other: Enhanced Usual Care — A standardized handout with information on what treatment options might be useful to start with based on EPDS score and stage of pregnancy or postpartum.
Other: MOVIN Care Platform — Virtual collaborative care intervention with a stepped care approach in which a care coordinator directs participants to one or more evidence-based virtual interventions as appropriate.
  Arms: MOVIN

SUMMARY:
Despite available treatments for perinatal mood disorders, only 20% of affected women receive treatment that results in remission of symptoms. In order to address gaps in equitable access to treatment the investigators developed the Reproductive Mental health of Ontario Virtual Intervention Network (MOVIN), a virtual collaborative care platform to optimize access for pregnant and postpartum people in Ontario. MOVIN combines collaborative and stepped-care approaches to treatment of perinatal depression and anxiety. The overall objective of this pilot randomized controlled trial (RCT) is to determine the feasibility of implementing a protocol for studying MOVIN for pregnant and postpartum individuals with significant symptoms of depression and anxiety (EPDS > 12) in order to inform the conduct of a larger scale evaluation. O will be randomized to either the MOVIN or control condition and will be asked to complete follow-up assessments 12- and 24-weeks post-randomization. Participants in the MOVIN arm will receive access to the MOVIN platform which includes a care coordinator to help them navigate various virtual treatments. Participants in the control condition will receive a resource list and will navigate the various options on their own.

DETAILED DESCRIPTION:
People with scores above 12 on the EPDS have a 10 times greater likelihood of having a diagnosis of depression than those with scores with 12 or less, so this is an appropriate cut-off. The primary endpoint is at 12 weeks post-randomization and the secondary endpoint is at 24 weeks post-randomization. Randomization will be performed as block randomization (varying block sizes) with a 1:1 allocation and will be stratified based on EPDS score (13-19 vs. 20 or greater). Participants who score 12 or less on the EPDS in their initial self-referral screen will be informed that they are not at high risk for having depressive or anxiety disorder and the current time, and can re-screen as needed. Participants whose score is in the 9-12 range (i.e. those who are not likely to be experiencing a depressive or anxiety disorder requiring mental health treatment, but might benefit from additional support) will receive an automated message that communicates their score and the acknowledgment of their possible need for support, and provides a list of resources in Ontario that may be helpful for them. These participants will be invited to re-screen at any time into the study, and will be asked permission to be re-contacted in future to determine which supports they used, if any.

ELIGIBILITY:
Inclusion criteria:

1. Residents of Ontario at least 18 years of age
2. Currently pregnant or mother* of a live infant 0-12 months of age living at the same residence *through natural birth, adoption or surrogacy, including cis women, non-binary and transgender people in all their diversity
3. EPDS > 12
4. Registered with a primary care provider

Exclusion criteria:

1. Experiencing active suicidal ideation (MINI International Neuropsychiatric Interview)
2. Active substance use disorder (GAIN-SS), current mania or psychosis (MINI Neuropsychiatric Interview)
3. Unable to access the internet or a device that can support the MOVIN platform
4. Unable to participate in English
5. Unable to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of the trial protocol: Recruitment | 12 weeks post randomization
  Measures of recruitment and retention include rate of recruitment, reason for non-participation and rate of completion of follow-up measures.
Feasibility of the trial protocol: Acceptability | 12 weeks post randomization
  Measures of acceptability include participants' overall experience and satisfaction with and acceptance of the MOVIN platform and the care coordinator, the care coordinator's assessment of the MOVIN platform and its impact on patient care, and primary care providers' assessment of MOVIN's impact on patient care.
Feasibility of the trial protocol: Compliance | 12 weeks post randomization
  Measures of compliance include rate of completion of MOVIN-specific activities, rate of completion of suggested interventions, and rate of resource use.

SECONDARY OUTCOMES:
Feasibility of the trial protocol: Recruitment | 24 weeks post randomization
  Measures of recruitment and retention include rate of recruitment, reason for non-participation and rate of completion of follow-up measures.
Feasibility of the trial protocol: Acceptability | 24 weeks post randomization
  Measures of acceptability include participants' overall experience and satisfaction with and acceptance of the MOVIN platform and the care coordinator, the care coordinator's assessment of the MOVIN platform and its impact on patient care, and primary care providers' assessment of MOVIN's impact on patient care.
Feasibility of the trial protocol: Compliance | 24 weeks post randomization
  Measures of compliance include rate of completion of MOVIN-specific activities, rate of completion of suggested interventions, and rate of resource use.
Maternal clinical outcomes - depression symptoms | 12 and 24 weeks post randomization
  Depressive symptoms will be measured using the Edinburgh Postnatal Depressive Scale (EPDS), a self-report scale that has been validated for use in pregnancy and postpartum. EPDS scores range from 0 to 30. EPDS scores >12 are predictive of a diagnosis of depression, with higher scores indicating more severe symptoms.
Maternal clinical outcomes - anxiety symptoms | 12 and 24 weeks post randomization
  Anxiety symptoms will be measured using the General Anxiety Disorder-7 (GAD-7) scale, which is a self-report scale with good discriminate validity in perinatal populations. GAD-7 scores range from 0 to 21, with higher scores indicating more severe symptoms.
Maternal clinical outcomes - quality of life | 12 and 24 weeks post randomization
  Quality of life will be measured using the 5 Level-5 Dimension EuroQol 5 (EQ-5D-5L) which is a multi-attribute utility instrument for measuring quality-adjusted life year (QALY), a preference-based utility measure of health-related quality of life as perceived by the patient. It can define 3125 different health states ranging from 11111 (full health) to 55555 (worst health).
Health service use: participant time | 12 and 24 weeks post randomization
  Measured by participant self-report of activities related to attending appointments and obtaining services.
Health service use: participant cost | 12 and 24 weeks post randomization
  Measured by participant self-report of costs related to attending appointments and obtaining services.
Health service use: health system costs | 12 and 24 weeks post randomization
  Calculated from participant self-report of medical costs such as hospitalizations, visits with health professionals and medications.
Care coordinator time | 12 and 24 weeks post randomization
  Care coordinator time per participant will be measured as the time spent per participant on the MOVIN platform, time spent on phone assessments and other related activities.
Care coordinator cost | 12 and 24 weeks post randomization
  Care coordinator cost per participant will be measured as the cost per participant on the MOVIN platform, on phone assessments and other related activities.
Dyadic relationship | 12 and 24 weeks post randomization
  The Dyadic Adjustment Scale (DAS) is a self-report measure of relationship adjustment with an intimate partner and will be used to measure relationship distress. The first 15 items of the 32-item measure will be used to assess dyadic consensus. Scores range fro 0 to 75. Higher scores indicate a higher degree of dyadic consensus.
Maternal child relationship | 12 and 24 weeks post randomization
  All participants who are postpartum at any time point will complete Parenting Stress Index short form (PSI-SF) to measure parenting stress. This is a 36-item measure consisting of 3 sub-scales: parental distress, dysfunction in the parent-child relations and difficult child. Scores range from 36 to 180. Higher scores indicate higher levels of parenting stress.
Infant temperament | Baseline, 12 and 24 weeks post randomization
  Infant temperament will be measured using the Infant Characteristics Questionnaire (ICQ), an instrument that assesses parental perceptions of difficult infant temperament. Scores range from 28 to 196. Higher scores indicate a higher level of parental perceptions of difficult infant temperament.

OTHER OUTCOMES:
Co-variates | Baseline
  We will collect sociodemographic, obstetrical and psychiatric history data. We will also conduct a diagnostic phone interview using the MINI International Neuropsychiatric Interview for major depressive disorder, obsessive-compulsive disorder, panic disorder, agoraphobia, social anxiety disorder, generalized anxiety disorder, alcohol and substance abuse, past (hypo)mania and psychosis, and post-traumatic stress disorder.
Maternal birth outcomes | Baseline, 12 and 24 weeks post randomization
  Self-reported pregnancy and birth complications, if applicable.
Neonatal birth outcomes | Baseline, 12 and 24 weeks post randomization
  Self-reported neonatal birth outcomes including medical conditions and complications, if applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Dalfen, MD, Principal Investigator — Women's College Hospital and Sinai Health System; Simone Vigod, MD, MSc, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada